CLINICAL TRIAL: NCT06387602
Title: Comparison Between Effects of Active Release Technique and Post Isometric Relaxation on Adductor Strain in Mixed Martial Arts Fighters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/6
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Adductor Strain
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ART Group (Experimental): Week 1 CRYOTHERAPY STRENGTHENING OF ADDUCTORS Adductor Isometrics Side-lying adductor strengthening Adductor resistance with stepper ACTIVE RELEASE TECHNIQUE Week 2 STRENGTHENING OF ADDUCTORS Adductor Isometrics Side-lying adductor strengthening Adductor resistance with stepper ACTIVE RELEASE TECHNIQUE
  Interventions: Procedure: Cryotherapy; Procedure: Strengthening of adductors; Procedure: Active release technique
- PIR Group (Experimental): Week 1 CRYOTHERAPY STRENGTHENING OF ADDUCTORS Adductor Isometrics Side-lying adductor strengthening Adductor resistance with stepper POST ISOMETRIC RELAXATION Week 2 STRENGTHENING OF ADDUCTORS Adductor Isometrics Side-lying adductor strengthening Adductor resistance with stepper POST ISOMETRIC RELAXATION
  Interventions: Procedure: Cryotherapy; Procedure: Strengthening of adductors; Procedure: Post-Isometric Relaxation

INTERVENTIONS:
Procedure: Cryotherapy — Take an icepack and wrap it in a moisture-absorbing towel. The temperature of the icepack should be between 1˚ to 10˚. Any temperature below 0˚ can damage the skin. The icepack will be on strained adductors for 5-7 minutes. Patients will be advised to do cryotherapy at home for 24-42 hours after every 2 hours.
Procedure: Strengthening of adductors — Both groups will perform the following strengthening of adductors which includes adductor isometrics, Side-lying adductor strengthening, and Adductor resistance with a stepper and will be done 10 repetitions, 3 times a week.
  After the performance of the Adductor strengthening protocol, Group A will be given the Active release technique while Group B will be given post-isometric relaxation by the therapist.
Procedure: Active release technique — Step 1: Place the body in a position (Dorsiflex ankle, flex the knee, extend the hip, flex the spine) so that the nerve is moved proximally. In this position, the nerve is relaxed on the distal side of the entrapment site and the nerve is tractioned on the proximal side.
  Step 2: Place contact between the distal Gracilis and the Sartorius and push the muscle proximally. The contact should not compress the nerve.
  Step 3: Move each joint so that the nerve moves distally past the muscle. The new position (Plantarflex and evert the ankle, extend the knee, flex the hip, extend the spine) will be achieved.
  Step 4: Move the contact to the proximal side of the muscles and push the muscle distally.
  Step 5: Move the nerve proximally again by pushing the muscle distally. This brings the position of the patient back to Step 1.
  Contact will be held for a short time 5-20 seconds with repetitions 3-5 times to the injury site and 2 sessions per week.
  Arms: ART Group
Procedure: Post-Isometric Relaxation — Step 1: Position the patient's limb at a point with the highest resistance felt during abduction.
  Step 2: The patient is asked to bring the leg back into adduction using only 20% of strength against firm resistance given by the therapist.
  Step 3: The patient will contract the agonist (the muscle that needs to be released) while holding an inhaled breath. Contraction should be held between 7-10 seconds without any jerking, bouncing, or wobbling.
  Step 4: The patient is asked to release their effort slowly and completely. As the patient relaxes, the limb is guided into a new resistance barrier where a bind is felt again.
  Step 5: After PIR, a 10-20-second latency period exists and the muscle can be stretched more easily.
  Contract adductor muscle for 7-10 seconds and relax the same for 7-10 seconds with repetitions 7 times and 2 sessions per week.
  Arms: PIR Group

SUMMARY:
This study is a randomized controlled trial and the purpose of this study is to compare the effects between active release technique and post-isometric relaxation on adductor strain in mixed martial arts fighters.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects between active release technique and post-isometric relaxation on adductor strain in mixed martial arts fighters on flexibility, pain, range of motion, and functionality, in adults (age: 20-35 years )

1. Numeric pain rating scale
2. Goniometer
3. Bent Knee Fall Out Test
4. Lower extremity functional scale Data will be collected before and after the intervention protocol for each participant.

Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Pre and post-intervention scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female genders
* Ages 20-35 years
* Professional Mixed Martial Arts fighters involved in kicking, sprinting, jumping, hiking
* Grade 1 or 2 adductor strain
* Clinical adductor dysfunction (pain reproduced by palpation of the enthesis, passive stretching of the adductors, and active resisted adduction)
* Numeric Pain Rating Scale (NPRS) 1-8
* Positive Bent Knee Fall Out (BKFO test)

Exclusion Criteria:

* Any clinical or radiographic evidence of pathological involvement of the hip joint (femoroacetabular impingement: pincer and/or cam features, dysplasia)
* Grade 3 adductor strain
* History of recent fracture

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 2 weeks
  Numeric Pain Rating Scale (NPRS): ICC (0.93-0.96) It has a scale of 0-10 or 0-100 points and can be given verbally or in writing.
Range of motion | 2 weeks
  It will be measured through goniometer
Functionality | 2 weeks
  It will be measured through lower extremity functional scale (LEFS)
Flexibility | 2 weeks
  It will be measured through bent knee fall out test

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan